CLINICAL TRIAL: NCT04139642
Title: Standing Balance as the Fifth Vital Sign in Clinical Setting
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Bertec Corporation (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ajit Chaudhari, Associate Professor of Physical Therapy, Orthopaedics, Mechanical Engineering, and Biomedical Engineering, Ohio State University
Other Study IDs: 2019H0265; R42AG062065-02 (NIH)
Record Dates: First submitted 2019-10-21; First posted 2019-10-25 (Actual); Results first posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-09

CONDITIONS: Accidental Fall; Postural Balance; Clinical Decision-making
Keywords: descriptive observational study; balance measurement

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group AB: A block randomization scheme by clinic type will be used to assign which clinics receive the Balance+Weight device in the first 9 months and which clinics receive the Balance+Weight device in the second 9 months. The block randomization scheme is proposed instead of simple randomization because of the expected variation between clinics in the types of patients they see. At the 9-month point, OSU personnel will go to every site to reprogram each device from Balance+Weight mode to Weight Only mode or vice versa, and to move the immediate feedback kiosks to the new Balance+Weight sites.
  Interventions: Device: SimpleSway
- Group BA: A block randomization scheme by clinic type will be used to assign which clinics receive the Balance+Weight device in the first 9 months and which clinics receive the Balance+Weight device in the second 9 months. The block randomization scheme is proposed instead of simple randomization because of the expected variation between clinics in the types of patients they see. At the 9-month point, OSU personnel will go to every site to reprogram each device from Balance+Weight mode to Weight Only mode or vice versa, and to move the immediate feedback kiosks to the new Balance+Weight sites.
  Interventions: Device: SimpleSway

INTERVENTIONS:
Device: SimpleSway — During the 9-month period each practitioner who receives the balance + weight device is asked to provide anonymous feedback via a kiosk regarding if the balance data influenced clinical decision making after every patient. The kiosk has four marked buttons indicating a 4-point Likert Scale, so the practitioner just presses one of the four buttons to indicate their agreement with the statement, "The balance measurement influenced my clinical decision making with this patient." After 9 months, the devices are switched so that every practitioner who had a weight only device receives balance + weight device and vice versa. After the second 9-month period concludes all devices will be retrieved by study personnel, and participants will be asked to complete surveys regarding their experience and attend group feedback sessions regarding their experiences.

SUMMARY:
This 18-month prospective, observational study involving real world data will determine if the use of a standing scale that delivers a quantitative measure of standing balance along with weight (balance + weight) in place of a scale that only delivers weight (weight only) influences clinical decision making by health care practitioners in the ambulatory outpatient setting. Providers will be randomized to receive the balance+weight scale or weight-only scale for 9 months, then to crossover and receive the other for 9 months. The primary outcome measures are (1) providers' self-reported perceptions of whether the balance measurement influences their clinical decision making and (2) the rate of performing falls risk assessments or referring to a specialist for evaluation and treatment based on aggregate billing data. The secondary outcome measure is qualitative interviews with practitioners regarding their perceptions on the utility and barriers to using the device.

DETAILED DESCRIPTION:
Recruitment of clinics to participate in study. Study personnel will recruit clinics to participate in an 18-month trial of the quantitative postural control assessment (Balance+Weight) device. Eligible clinics include any that self-report a substantial component of their patient population that may be at risk of falls, but that are not a referral site for patients previously identified as being at elevated falls risk. In clinics where multiple providers see patients, at least one provider must be willing to participate and commit to placing the novel device in their clinic, as well as to the other components of participation detailed below. Due to the number of ambulatory care clinics within a radius to allow same-day servicing of the devices and resource limitations to manufacture units, the investigators will cap recruitment when the investigators reach 20 clinics or 60 devices in service, whichever is reached first. Every participating clinic will have the opportunity to receive the device that delivers Balance+Weight either immediately or after a 9-month waiting period depending on randomization.

Randomization of clinics. A block randomization scheme by clinic type will be used to assign which clinics receive the Balance+Weight device in the first 9 months and which clinics receive the Balance+Weight device in the second 9 months. The block randomization scheme is proposed instead of simple randomization because of the expected variation between clinics in the types of patients they see. Blocks will be determined based on the estimated percent of patients seen who are over 65, diabetic, undergoing chemotherapy (all oncology clinics), or are using assistive devices during some of their care (e.g. orthopaedic trauma clinics). Clinics for whom 50% or more of their patients are in any of these categories will be included in one block, whereas clinics for whom less than 50% of their patients are in any of these categories will be included in the other block. While this scheme does not fully account for the confounder of multiple risk factors for falls or multiple co-morbidities in some clinics, equipoise between treatment arms is also achieved through the crossover design whereby every clinic serves as its own control as well.

Training of clinics. At delivery of the Balance+Weight device to the clinic, a one-hour in-service will be performed by study personnel to train all providers and medical assistants on its proper use and the entry of data into the electronic medical record. This training will include how to operate the device and how to use the accompanying documentation with the reported data to inform clinical decision-making. This documentation will include threshold values for likelihood of the patient's balance being Within Normal Limits as well as the change in value that would indicate a change in the patient's balance status along with appendices that contain the published peer-reviewed journal articles upon which these recommendations are based. Upon request by the clinic, study personnel will repeat the training if refreshers are needed by clinic staff. An unlimited number of refresher trainings are permitted for each clinic, and the number of trainings requested per clinic will be recorded.

Incorporation of quantitative postural control assessment device into clinic flow including immediate feedback on clinical utility. Each participating clinic will place the study device in a location to allow its use instead of their weight scale. In the Balance+Weight arm, the device is capable of either just giving weight, or of providing balance data if the patient stands quietly with eyes closed for 30s. In the Weight Only arm, the device only gives a weight measurement, just as a standard weight scale would. In both cases, the provider and their staff make their own clinical decisions as to which patients to make measurements of and how to use the provided information. The medical assistant may choose to enter the appropriate values into the medical record and continue with any other standard procedures in that clinic setting as part of the rooming or initial evaluation process. The provider can then examine the recorded balance measurement along with their standard examination and determine whether any further evaluations in that clinic or referral to a specialist, physical therapy, or other falls prevention is appropriate and record that diagnosis or referral into the medical record.

Immediate feedback from provider on clinical decision-making process. After each patient encounter in which the provider assessed balance using the Balance+Weight device, the provider who made a clinical decision regarding balance or falls risk is asked to press a button on a small kiosk that the investigators will provide which logs their agreement with the statement, "The balance measurement influenced my clinical decision making with this patient." These kiosks from Happy-Or-Not.com are completely wireless and use their own 3G network to communicate the results of a single 4-point Likert scale question back to a central server that the study staff can monitor to collect data and get a real-time indication of whether the providers are using the Balance+Weight device.

Crossover of sites after 9 months. At the 9-month point, study personnel will go to every site to reprogram each device from Balance+Weight mode to Weight Only mode or vice versa, and to move the immediate feedback kiosks to the new Balance+Weight sites.

Data pull of clinic-level diagnosis and referral data. At or just after the crossover between sites has occurred, study personnel in conjunction with the IT departments at participating sites will pull the clinic diagnosis and referral data for all participating providers. After Casey et al.[1], our initial plan is to count instances of the following Common Procedural Terminology (CPT) Category II codes:

(Primary) CPT II 3288: Assessment of falls risk CPT II 0518: Development of a falls care plan CPT II 1101: Documentation of falls in past year (no falls/ single fall without injury) CPT II 1100: Documentation of an injurious fall/ multiple falls Other referral codes as appropriate Because CPT codes are updated each calendar year, the investigators will review the new codes each year and revise this code list as new codes related to falls assessment are added or subtracted. The investigators will pull this data from both the 9 months of participation in the study, as well as the same 9 month period in the calendar year before the study began as a historical control. The data will be pulled again upon completion of the study for the second 9-month period.

Focus group discussions after completion of RCT. Following conclusion of the trial, The investigators will engage all participants in focus groups regarding their experience using the Balance+Weight device. These discussions are intended to complement and enrich our understanding of how the users of the device (providers and medical assistants) either benefitted or did not benefit from having it in the clinic. Feedback will be used to assess the implementation toolkit and inform the development of the final version of the toolkit. Seed questions for these focus groups include:

In what ways, if any, did participants find having a quantitative postural control assessment on every patient useful in their clinical decision making? If participants applied the device's data differently for different patients, how did participants use it across these different patients? Did the time it took to make the measurement or interpret the measurement impact the efficiency of their clinic (positively or negatively) and how? In what ways could the investigators better implement and train participants to use the device, and use it with the electronic medical record?

ELIGIBILITY:
Inclusion Criteria:

* Columbus Metropolitan Area by the following counties: Franklin, Madison, Union, Delaware, Locking, Fairfield, Pickaway.
* Physician, advanced practice registered nurse, or physician assistant, who diagnoses and treats patients in ambulatory outpatient settings
* self-report that falls are a concern for a significant fraction of the participant's patients, where the participants defines significant as they see fit.
* Participants must commit to using the test device as the primary weight scale in the clinic for the duration of the study to be selected.

Exclusion Criteria:

* No gender, ethnic, or racial groups will be excluded from this study, though it is expected that the majority of the sample will be Caucasian American, given that the professions of physicians, nurse practitioners, and physician assistants are predominantly Caucasian American.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will include physicians, advanced practice registered nurses, and physician assistants who diagnose and treat patients in ambulatory outpatient settings. Participants must commit to using the test device as the primary weight scale in the clinic for the duration of the study to be selected. Participants will be identified through word-of-mouth and email announcements distributed by the organizations listed above. Any additional organizations that express interest will also be encouraged to distribute announcements to their employees.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Result] Casey CM, Parker EM, Winkler G, Liu X, Lambert GH, Eckstrom E. Lessons Learned From Implementing CDC's STEADI Falls Prevention Algorithm in Primary Care. Gerontologist. 2017 Aug;57(4):787-796. doi: 10.1093/geront/gnw074. Epub 2016 Apr 29. PMID 27130270

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible clinics include any in the Columbus Ohio Metropolitan Area that self-report a substantial component of their patient population that may be at risk of falls, but that are not a referral site for patients previously identified as being at elevated falls risk. The investigators planned to cap recruitment when the investigators reach 20 clinics or 60 devices in service, whichever is reached first.
Pre-assignment Details: A total of 3 participants were never assigned. Of these excluded particpants, 2 were lost to follow-up and 1 never received the intervention device due to moving to a different clinic and not notifying the study.
Units Other Than Participants: clinics
Groups:
- Group AB; Group BA: A block randomization scheme by clinic type will be used to assign which clinics receive the Balance+Weight device in the first 9 months (AB) and which clinics receive the Balance+Weight device in the second 9 months (BA). The block randomization scheme is proposed instead of simple randomization because of the expected variation between clinics in the types of patients they see. At the 9-month point, OSU personnel will go to every site to reprogram each device from Balance+Weight mode to Weight Only mode or vice versa, and to move the immediate feedback kiosks to the new Balance+Weight sites. The historical control time period for all participants includes a 12-month period before the beginning of the first intervention, from March 2019-February 2020. The first intervention period went from November 2020-July 2021, and the second intervention period went from August 2021-April 2022.
  SimpleSway: During 9-month A period participants provide anonymous feedback via a kiosk with four marked buttons indicating a 4-point Likert Scale. Participant presses button to indicate agreement with statement, "The balance measurement influenced my clinical decision making with this patient." After 9 months, the devices are switched so that every practitioner who had a weight only device receives balance + weight device and vice versa. After second 9-month period all devices are retrieved, and participants complete surveys and attend group feedback sessions regarding their experiences.
Period: Historical Control Period (12 Months)
Arm/Group | Group AB | Group BA
Started | 20; 8 clinics | 22; 8 clinics
Completed | 20; 8 clinics | 22; 8 clinics
Not Completed | 0; 0 clinics | 0; 0 clinics
Period: First Intervention (9 Months)
Arm/Group | Group AB | Group BA
Started | 20; 8 clinics | 22; 8 clinics
Completed | 20; 8 clinics | 21; 7 clinics
Not Completed | 0; 0 clinics | 1; 1 clinics
Not completed — Permission denied to use the device by clinic manager | 0 | 1
Period: Second Intervention (9 Months)
Arm/Group | Group AB | Group BA
Started | 20; 8 clinics | 21; 7 clinics
Completed | 20; 8 clinics | 21; 7 clinics
Not Completed | 0; 0 clinics | 0; 0 clinics

BASELINE CHARACTERISTICS:
Population: Providers whose patient populations include a significant number of people considered by the provider to be at risk of falls. The populations of Groups AB and BA only include participants who were assigned to a group and who received a device in the first intervention period.
Groups:
- Group AB: Participants who received the Balance+Weight device during the First Intervention Period (9 months), then the Weight Only device during the Second Intervention Period (9 months).
- Group BA: Participants who received the Weight Only device during the First Intervention Period (9 months), then the Balance+Weight device during the Second Intervention Period (9 months).
- Total: Total of all reporting groups
Arm/Group | Group AB | Group BA | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 21 | 41
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender - Biological Sex is not relevant because these were health care providers and the study was investigating their clinical decision-making.
  Participants
    Man | 12 | 8 | 20
    Woman | 8 | 13 | 21
    Gender-Fluid or Non-Binary | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Degree or Credential [Count of Participants; unit: Participants]
  Medical Doctor | 20 | 14 | 34
  Doctor of Osteopathy | 0 | 3 | 3
  Certified Nurse Practitioner | 0 | 3 | 3
  Physician Assistant | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Balance-Related Diagnoses
Description: Percent of unique visits with a balance-related diagnosis
Time Frame: Historical control period plus 18-month intervention period
Population: All unique in-person visits by patients to the providers who participated in the study
Measure: Count of Units; unit: unique visits
Units Other Than Participants: unique visits
Groups:
- A: Balance+Weight: Participants during the 9-month that they had the Balance+Weight device available in their clinic.
- B: Weight-Only: Participants during the 9-month period when they had a device that only reports weight.
- Historical Control: Participants during the historical period March 2019-February 2020 before the intervention began
Arm/Group | A: Balance+Weight | B: Weight-Only | Historical Control
Number analyzed (Participants) | 41 | 41 | 41
Number analyzed (unique visits) | 41726 | 38236 | 69224
unique visits | 12118 | 11763 | 19904
Statistical Analysis 1: Comparison: A: Balance+Weight vs B: Weight-Only vs Historical Control; The null hypothesis was that the rate of balance-related diagnosis as a percentage of total visits would be the same between the historical control period, the active control (weight-only), and the intervention (balance+weight), considering provider and month as co-variates; Test type: Superiority; p < 0.0001, Mixed Models Analysis — A mixed-effects model with provider as a random effect and month as a fixed effect was used to test the main effect of arm

2. Primary Outcome: Number of Unique Visits With and Without Balance-Related Referrals
Description: Difference in the rate of performing falls risk assessments or referring to a specialist for evaluation and treatment based on aggregate billing data when the provider has the device versus when the provider does not have the device.
Time Frame: at conclusion of second intervention period (18 months)
Population: Physicians and advanced-practice providers who were granted access to the intervention device to use with their patients according to their clinical judgment.
Measure: Count of Units; unit: unique visits
Units Other Than Participants: unique visits
Arm/Group | A: Balance+Weight | B: Weight-Only | Historical Control
Number analyzed (Participants) | 41 | 41 | 41
Number analyzed (unique visits) | 41726 | 38236 | 69224
unique visits
  visits with balance-related referral | 474 | 479 | 1145
  visits without balance-related referral | 41252 | 37757 | 68079
Statistical Analysis 1: Comparison: A: Balance+Weight vs B: Weight-Only vs Historical Control; The null hypothesis was that the rate of balance-related referral as a percentage of total visits would be the same between the historical control period, the active control (weight-only), and the intervention (balance+weight), considering provider and month as co-variates; Test type: Superiority; p = 0.15, Mixed Models Analysis — Mixed-effects model with provider as a random effect and month as a fixed effect. Statistical significance a priori threshold set at 0.05

3. Primary Outcome: Providers' Perceptions Reported as Number of Responses
Description: Providers' self-reported perceptions of whether the balance measurement influences their clinical decision making.
Time Frame: through study completion, an average of 18 months
Population: During the time in which they had a balance device (intervention A), all participants had access to a device that would record an instantaneous momentary assessment of their agreement with the statement, "The balance device influenced my clinical decision-making today." The statement is irrelevant when a balance device was not present, so this outcome only is collected when they had the Balance+Weight device, regardless of group assignment.
Measure: Number; unit: responses
Units Other Than Participants: Responses
Groups:
- Group AB: Participants who had the Balance+Weight device present and available in their clinic during the First Intervention Period.
- Group BA: Participants who had the Balance+Weight device present and available for use in their clinic during the Second Intervention Period.
Arm/Group | Group AB | Group BA
Number analyzed (Participants) | 20 | 21
Number analyzed (Responses) | 361 | 1073
responses
  Very Positive | 117 | 347
  Somewhat Positive | 115 | 455
  Somewhat Negative | 47 | 226
  Very Negative | 82 | 45

ADVERSE EVENTS:
Time Frame: 18 months
Groups:
- Balance+Weight; Weight Only: A block randomization scheme by clinic type will be used to assign which clinics receive the Balance+Weight device in the first 9 months and which clinics receive the Balance+Weight device in the second 9 months. The block randomization scheme is proposed instead of simple randomization because of the expected variation between clinics in the types of patients they see. At the 9-month point, OSU personnel will go to every site to reprogram each device from Balance+Weight mode to Weight Only mode or vice versa, and to move the immediate feedback kiosks to the new Balance+Weight sites.
  SimpleSway: During the 9-month period each practitioner who receives the balance + weight device is asked to provide anonymous feedback via a kiosk regarding if the balance data influenced clinical decision making after every patient. The kiosk has four marked buttons indicating a 4-point Likert Scale, so the practitioner just presses one of the four buttons to indicate their agreement with the statement, "The balance measurement influenced my clinical decision making with this patient." After 9 months, the devices are switched so that every practitioner who had a weight only device receives balance + weight device and vice versa. After the second 9-month period concludes all devices will be retrieved by study personnel, and participants will be asked to complete surveys regarding their experience and attend group feedback sessions regarding their experiences.
Arm/Group | Balance+Weight | Weight Only
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 0/41

LIMITATIONS AND CAVEATS:
Intervention was likely affected by the COVID-19 pandemic affecting both volume and characteristics of the patients visiting the clinics of the providers who participated in the study. Several provider participants noted in post-intervention focus groups that they were unable to implement the intervention device into their clinical workflow due to pandemic-related workforce shortages and turnover.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/42/NCT04139642/Prot_SAP_001.pdf